CLINICAL TRIAL: NCT02371616
Title: A Clinical Study to Evaluate the Efficacy of Two Dentifrices for Dentine Hypersensitivity
Brief Title: Clinical Study to Evaluate the Efficacy of Two Dentifrices for Dentine Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202199
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2017-12

CONDITIONS: Dentine Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Sodium Fluoride; fluorophosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test dentifrice (Experimental): Test dentifrice containing 5% w/w calcium sodium phosphosilicate and 1426 ppm fluoride as sodium flouride
  Interventions: Device: Calcium sodium phosphosilicate; Other: Sodium fluoride
- Comparator dentifrice (Active Comparator): Comparator dentifrice containing 5% w/w calcium sodium phosphosilicate and 1426 ppm fluoride as sodium monofluorophosphate
  Interventions: Device: Calcium sodium phosphosilicate; Other: Sodium monofluorophosphate

INTERVENTIONS:
Device: Calcium sodium phosphosilicate — 5% w/w calcium sodium phosphosilicate
Other: Sodium fluoride — 1426 ppm fluoride as sodium fluoride
  Arms: Test dentifrice
Other: Sodium monofluorophosphate — 1426 ppm fluoride as sodium monofluorophosphate
  Arms: Comparator dentifrice

SUMMARY:
An 8 week clinical study to evaluate the ability of an experimental dentifrice containing calcium sodium phosphosilicate and sodium fluoride to provide relief from dentine hypersensitivity compared to a marketed dentifrice containing calcium sodium phosphosilicate and sodium monofluorophosphate.

DETAILED DESCRIPTION:
A single centre, multi-site, randomised, examiner blind, two treatment, parallel group, non-inferiority design clinical study conducted in healthy subjects with self-reported and clinically diagnosed dentine hypersensitivity (DH). This study will compare the effectiveness of a test dentifrice containing 5% w/w calcium sodium phosphosilicate and fluoride as sodium fluoride to a commercially available dentifrice containing 5% w/w calcium sodium phosphosilicate and fluoride as sodium monofluorophosphate, in providing relief from DH after 4 and 8 weeks twice daily treatment.

ELIGIBILITY:
Inclusion Criteria:

* subjects in good general health with no clinically significant/ relevant abnormalities of oral examination
* pre-existing self reported and clinically diagnosed tooth sensitivity
* at screening a minimum of 20 natural teeth and at least two accessible, non-adjacent teeth (incisors, canines or pre-molars) with signs of erosion or abrasion and/or facial/cervical gingival recession (EAR), with a Gingival Index ≤1 and clinical mobility ≤1, and with signs of DH as measured by qualifying evaporative (air) assessment
* at baseline, a minimum of 2 non-adjacent accessible teeth (incisors, canines or premolars) with DH (qualifying tactile threshold Yeaple ≤ 20g, Schiff Sensitivity Score ≥ 2)

Exclusion Criteria:

* subjects with a known or suspected intolerance or hypersensitivity to study products
* presence of chronic debilitating disease which could affect study outcomes
* any condition which is causing dry mouth
* use of an oral care product indicated for the relief of dentine hypersensitivity
* participation in a DH treatment study in the 8 weeks prior to screening
* taking daily doses of a medication/ treatment which could interfere with perception of pain or is causing dry mouth
* require antibiotic prophylaxis for dental procedures
* dental prophylaxis within 4 weeks of screening
* treatment of periodontal disease within 12 months of screening+C60
* scaling or root planing within 3 months of screening
* tooth bleaching within 8 weeks of screening
* active caries or periodontitis
* partial dentures, orthodontic appliances or dental implants which could affect study outcomes
* Pregnant and breast-feeding females
* Main Exclusions for Test Teeth: evidence of current or recent caries; treatment of decay within 12 months of screening; teeth with exposed dentine but with deep, defective or facial restorations; teeth used as abutments for fixed or removable partial dentures; teeth with full crowns or veneers, orthodontic bands or cracked enamel; sensitive teeth with contributing aetiologies other than erosion, abrasion or recession

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 304 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2014-12-18 (Actual); Study Completion 2014-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Ellesmere Port, Cheshire
  - GSK Investigational Site, Maldon, Essex
  - GSK Investigational Site, Metropolitan Borough of Wirral

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center (three sites) in United Kingdom.
Pre-assignment Details: A total of 731 participants were screened, out of which 304 participants were randomized. 427 participants were not randomized because 377 did not met the study criteria, 1 had adverse event, 3 were lost to follow up and 1 due to protocol violation, 5 withdrew consent and 40 participants were not randomized because of other reasons (not specified).
Groups:
- Test Dentifrice: Test dentifrice containing 5% weight by weight (w/w) calcium sodium phosphosilicate and 1426 parts per million (ppm) fluoride as sodium fluoride.
Period: Overall Study
Arm/Group | Test Dentifrice | Comparator Dentifrice
Started | 150 | 154
Completed | 146 | 147
Not Completed | 4 | 7
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal of Consent | 1 | 0
Not completed — Other (Not specified) | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Test Dentifrice: Test dentifrice containing 5% w/w calcium sodium phosphosilicate and 1426 ppm fluoride as sodium fluoride.
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice | Comparator Dentifrice | Total
Number analyzed (Participants) | 150 | 154 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.33) | 42.5 (9.43) | 41.9 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 131 | 253
  Male | 28 | 23 | 51

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Evaporative Air Sensitivity as Measured by Visual Analogue Score (VAS) at Week 8
Description: Evaporative air sensitivity was assessed by examiner as a response to a 1 second application of air from a triple air dental syringe applied to the exposed dentine surface of hypersensitive tooth from a distance of approximately 1centimeter. Each participants rated the intensity of their response to the stimulus using a 100 millimeter (mm) VAS, were 0 represented "no pain" and 100 represented the" worst pain imaginable". Change from baseline was calculated as mean score at the given time point minus mean score at baseline of the two selected test teeth.
Time Frame: At Baseline and Week 8
Population: Analysis for this outcome was performed on per protocol (PP) population which is defined as all participants in the intent to treat (ITT) population who had at least one assessment of efficacy considered unaffected by protocol violations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice | Comparator Dentifrice
Number analyzed (Participants) | 147 | 149
score on a scale
  At Baseline | 53.05 (20.873) | 55.89 (21.334)
  At Week 8: number analyzed (Participants) | 146 | 144
  At Week 8 | 31.62 (24.194) | 30.51 (23.960)
  Change from baseline at Week 8: number analyzed (Participants) | 146 | 144
  Change from baseline at Week 8 | -21.50 (22.231) | -25.16 (22.322)
Statistical Analysis 1: Comparison: Test Dentifrice vs Comparator Dentifrice; Statistical analysis applies to change from baseline at week 8 for test and comparator dentifrice; Test type: Non-Inferiority — Inferences: upper end of the 2-sided 95% CI for the treatment difference for the estimated effect of Test relative to Comparator, for success, should be <=6mm. (i.e., Test is no more than 6mm inferior to Comparator); p = 0.2678, ANCOVA — From ANCOVA model: change from baseline as the response variable, treatment group, baseline Schiff stratum and study site as fixed effects, with baseline VAS score as covariate; Least square (LS) mean difference = 2.67, 95% CI 2-sided [-2.06 to 7.40] — Difference is first named treatment minus second named dentifrice such that a negative difference favors the first named treatment

2. Secondary Outcome: Mean Change From Baseline in Evaporative Air Sensitivity as Measured by Visual Analogue Score (VAS) at Week 4
Description: Evaporative air sensitivity was assessed by examiner as a response to a 1 second application of air from a triple air dental syringe applied to the exposed dentine surface of hypersensitive tooth from a distance of approximately 1centimeter. Each participants rated the intensity of their response to the stimulus using a 100 mm VAS, were 0 represented "no pain" and 100 represented the" worst pain imaginable". Change from baseline was calculated as mean score at the given time point minus mean score at baseline of the two selected test teeth.
Time Frame: At Baseline and Week 4
Population: Analysis for this outcome was performed on PP population which is defined as all participants in the ITT population who had at least one assessment of efficacy considered unaffected by protocol violations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice | Comparator Dentifrice
Number analyzed (Participants) | 147 | 149
score on a scale
  At Week 4: number analyzed (Participants) | 145 | 148
  At Week 4 | 40.71 (22.828) | 40.60 (23.090)
  Change from baseline at Week 4: number analyzed (Participants) | 145 | 148
  Change from baseline at Week 4 | -12.12 (18.438) | -15.24 (19.895)

3. Secondary Outcome: Mean Change From Baseline in Evaporative Air Sensitivity as Measured by Schiff Sensitivity Score at Week 4 and Week 8
Description: Evaporative air sensitivity was measured by examiner as the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicate improvement in sensitivity. Change from baseline was calculated as mean score at the given time point minus mean score at baseline of the two selected test teeth.
Time Frame: At Baseline, Week 4 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Dentifrice | Comparator Dentifrice
Number analyzed (Participants) | 147 | 149
score on a scale
  At Baseline | 2.72 (0.393) | 2.68 (0.400)
  At Week 4: number analyzed (Participants) | 145 | 148
  At Week 4 | 2.13 (0.771) | 2.11 (0.832)
  Change from baseline at Week 4: number analyzed (Participants) | 145 | 148
  Change from baseline at Week 4 | -0.59 (0.689) | -0.57 (0.745)
  At Week 8: number analyzed (Participants) | 146 | 144
  At Week 8 | 1.65 (0.990) | 1.58 (1.002)
  Change from baseline at Week 8: number analyzed (Participants) | 146 | 144
  Change from baseline at Week 8 | -1.08 (0.922) | -1.09 (0.937)

4. Secondary Outcome: Change From Baseline in Tactile Threshold at Week 4 and Week 8
Description: Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentine surface from 10 g to an upper threshold of 80g in increments of 10 g. The tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. Change from baseline was calculated as mean score at the given time point minus mean score at baseline of the two selected test teeth.
Time Frame: At Baseline, Week 4 and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | Test Dentifrice | Comparator Dentifrice
Number analyzed (Participants) | 147 | 149
gram (g)
  At Baseline | 12.79 (3.419) | 12.18 (2.982)
  At Week 4: number analyzed (Participants) | 145 | 148
  At Week 4 | 25.45 (20.573) | 23.61 (18.616)
  Change from baseline at Week 4: number analyzed (Participants) | 145 | 148
  Change from baseline at Week 4 | 12.72 (20.181) | 11.42 (18.099)
  At Week 8: number analyzed (Participants) | 146 | 144
  At Week 8 | 32.88 (25.392) | 33.58 (24.840)
  Change from baseline at Week 8: number analyzed (Participants) | 146 | 144
  Change from baseline at Week 8 | 20.10 (25.041) | 21.42 (24.450)

ADVERSE EVENTS:
Arm/Group | Test Dentifrice | Comparator Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/154
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/154
Other Adverse Events (participants affected / at risk) | 51/150 | 59/154
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (N=150) | Comparator Dentifrice (N=154)
Rhinitis (Infections and infestations) | 9 | 12
Oral Herpes (Infections and infestations) | 7 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 6
Influenza (Infections and infestations) | 2 | 1
Tonsillitis (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
Ear Infection (Infections and infestations) | 0 | 1
Eye Infection (Infections and infestations) | 0 | 1
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 1 | 0
Toothache (Gastrointestinal disorders) | 4 | 5
Chapped Lips (Gastrointestinal disorders) | 1 | 3
Aphthous Stomatitis (Gastrointestinal disorders) | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 3
Cheilitis (Gastrointestinal disorders) | 1 | 1
Gingival Pain (Gastrointestinal disorders) | 1 | 1
Lip Ulceration (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Oral discomfort (Gastrointestinal disorders) | 0 | 2
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Oral Mucosal Exfoliation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Oral Disorder (Gastrointestinal disorders) | 0 | 1
Oral Mucosal Erythema (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1
Tongue Discolouration (Gastrointestinal disorders) | 0 | 1
Tongue Ulceration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 16 | 8
Migraine (Nervous system disorders) | 0 | 1
Lip Injury (Injury, poisoning and procedural complications) | 2 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 3 | 1
Mouth injury (Injury, poisoning and procedural complications) | 2 | 1
Traumatic Ulcer (Injury, poisoning and procedural complications) | 1 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Device Failure (General disorders) | 2 | 5
Application Site Discomfort (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.